CLINICAL TRIAL: NCT00000838
Title: A Phase II, Randomized Study of the Antiviral Activity and Resistance Interactions of Lamivudine (3TC) in Combination With Zidovudine (AZT), Stavudine (d4T), or Didanosine (ddI) Versus Monotherapy With ddI or d4T in HIV-Infected Individuals With 200 - 600 CD4+ Cells/mm3 and No Previous Nucleoside Experience
Brief Title: Antiviral Activity of and Resistance to Lamivudine in Combination With Zidovudine, Stavudine, or Didanosine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 306; 11281 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; Stavudine; Lamivudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To evaluate the efficacy, safety, and pharmacokinetics of lamivudine (3TC) combined with zidovudine (AZT), stavudine (d4T), or didanosine (ddI) in comparison with d4T or ddI monotherapy in HIV-infected patients with no prior nucleoside therapy.

3TC may be uniquely effective in combination with AZT due to the interaction of AZT and 3TC resistance mutations. One explanation is that the M184V mutation, which confers resistance to 3TC, suppresses AZT resistance. This benefit of 3TC may not extend to combination therapy with other nucleoside analogs.

DETAILED DESCRIPTION:
3TC may be uniquely effective in combination with AZT due to the interaction of AZT and 3TC resistance mutations. One explanation is that the M184V mutation, which confers resistance to 3TC, suppresses AZT resistance. This benefit of 3TC may not extend to combination therapy with other nucleoside analogs.

Patients are randomized to either a ddI limb or d4T limb, then randomized a second time to one of six treatment arms, as follows: ddI alone, d4T alone, 3TC/AZT (on both ddI and d4T limbs), 3TC/ddI, and 3TC/d4T. Treatment is given for 48 weeks. At study week 24, patients on monotherapy will have 3TC added to their regimen (in a blinded fashion).

PER AMENDMENT 10/18/96: A treatment extension phase has been added to the study design in order to allow subjects who complete 48 weeks of therapy to remain on their same blinded treatment until approximately 2 months after the last enrolled subject completes 48 weeks on the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis.

Patients must have:

* HIV infection.
* CD4 count 200 - 600 cells/mm3.
* Life expectancy of at least 24 weeks.
* Consent of parent or guardian if less than 18 years old.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Unexplained temperature >= 38.5 C for 7 consecutive days within 30 days prior to study entry.

PER AMENDMENT 1/25/96:

* A malignancy that requires systemic chemotherapies other than Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Concurrent other antiretroviral or immunologic agents.
* Other experimental therapies.
* Systemic corticosteroids (except as adjuvant therapy for acute PCP) and other immunosuppressive drugs.
* Systemic cytotoxic chemotherapy.
* Induction or maintenance with foscarnet or ganciclovir (oral or IV).

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* History of grade 2 or higher peripheral neuropathy.

Prior Medication:

Excluded:

* Antiretrovirals within 90 days prior to study entry.
* More than 7 days total lifetime use of any antiretroviral nucleoside.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256
Dates: Study Completion 1998-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuritzkes D, Study Chair; Johnson V, Study Chair
Locations (32):
- United States (31):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Marschner I, Betensky RA, Degruttola V, Kuritzkes DR. Biases in the assessment of viral load reduction in HIV clinical trials. Int Conf AIDS. 1998;12:802 (abstract no 42149)
- [Background] Hill A, Demasi R, Kuhn M. Different analyses give highly variable estimates of HIV-1 RNA undetectability and log reduction in clinical trials. Int Conf AIDS. 1998;12:813-4 (abstract no 42204)
- [Background] Kuritzkes DR, Marschner IC, Johnson VA, Bassett RL, Eron JJ, Fischl MA, Boone G, Skovronski J, Wood K, Bell DL, Pettinelli CB, Sommadossi JP. A randomized, double-blind, placebo-controlled trial of lamivudine (3TC) in combination with zidovudine (ZDV), stavudine (d4T), or didanosine (ddI) in treatment naive patients. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:79 (abstract no 1)
- [Background] Kuritzkes DR, Marschner I, Johnson VA, Bassett R, Eron JJ, Fischl MA, Murphy RL, Fife K, Maenza J, Rosandich ME, Bell D, Wood K, Sommadossi JP, Pettinelli C. Lamivudine in combination with zidovudine, stavudine, or didanosine in patients with HIV-1 infection. A randomized, double-blind, placebo-controlled trial. National Institute of Allergy and Infectious Disease AIDS Clinical Trials Group Protocol 306 Investigators. AIDS. 1999 Apr 16;13(6):685-94. doi: 10.1097/00002030-199904160-00009. PMID 10397563
- [Background] Kuritzkes DR, Bassett RL, Hazelwood JD, Barrett H, Rhodes RA, Young RK, Johnson VA; Adult ACTG Protocol 306 370 Teams. Rate of thymidine analogue resistance mutation accumulation with zidovudine- or stavudine-based regimens. J Acquir Immune Defic Syndr. 2004 May 1;36(1):600-3. doi: 10.1097/00126334-200405010-00008. PMID 15097303
- [Background] Fisher M. Nucleoside combinations for antiretroviral therapy: efficacy of stavudine in combination with either didanosine or lamivudine. AIDS. 1998;12 Suppl 3:S9-16. PMID 15168718